## Effects of Music-Based Occupational Therapy Activities on Attention Executive Functions in Children with Attention Deficit and Hyperactivity Disorder

15.04.2022

## INFORMED VOLUNTARY CONSENT FORM

It is known that sensory systems in early life have an important impact on the child's development and contribute to the development of cognitive and behavioral processes such as attention, as well as learning skills. In this context, possible problems in the registration and organization of sensory stimuli require comprehensive assessment and intervention. Within the scope of the occupational therapy services provided for the pediatric population at Istanbul Medipol University, Department of Occupational Therapy, the current health status of children applying for services is comprehensively evaluated in terms of physical, psychological, social, and environmental aspects. In areas requiring intervention, treatment goals and plans are determined collaboratively with parents through shared goal setting. Receiving the provided service is entirely voluntary. You have the right to refuse the service or discontinue participation at any time. In either case, there will be no penalty or loss of entitled benefits. If you agree to receive the service, no additional fee will be requested from you or from the institution providing your social security. The assessments and interventions to be conducted do not contain any risks.

The data obtained from this service will be used solely for research and educational purposes, and your personal identity information will remain strictly confidential. If you agree to participate, this form will be completed and signed by you and Occupational Therapist İbrahim Erarslan, and a copy will be given to you for your records. I have read the purpose and method of the service described above, had the opportunity to ask questions and discuss them, and received satisfactory answers. I was verbally informed about the possible risks and benefits of the service. I understand that I am receiving this service voluntarily, that I may withdraw at any time with or without reason, and that my current condition will not be adversely affected if I withdraw.

Under these conditions, I voluntarily agree to receive the mentioned service without any pressure or coercion (for myself / for my child / for my dependent).

If necessary, I consent to the access of my personal information by the specified person/institution/organization, and I also give permission for the data obtained from the service to be used for publication, archiving, or—if needed—transferred abroad for scientific contribution, provided that my identity information remains confidential.

Participant's Full Name:

Caregiver's Full Name: Service Provider's Full Name: Occupational Therapist İbrahim ERARSLAN